CLINICAL TRIAL: NCT03290807
Title: The Role of Tc 99m MDP SPECT/CT in Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma El-Zahraa Mostafa Mahmoud, resident physicians, Assiut University
Other Study IDs: SPECT/CT in osteoarthritis
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SPECT/CT — Combined single photon emission computerized tomography and conventional computerized tomography (SPECT/CT) is a hybrid imaging modality, which combines a 3D bone scintigraphy (SPECT) and a conventional CT into one imaging procedure. The use of SPECT/CT offers the benefit of combined anatomical, mechanical (CT) and functional imaging (SPECT)

SUMMARY:
Evaluation of the diagnostic value of SPECT/CT in patients with knee and/or hip OA, whether it is related to clinical findings and it could reflect clinical disease activity, and to determine the usefulness of SPECT/CT in early detection of OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a slowly developing chronic degenerative joint disease that progresses over years. After the classification and reporting of OA were established by American College of Rheumatology in 1986, the diagnosis has depended on the patients' symptoms and supported by plain radiographic findings.

Since X-ray image has a discrepancy with clinical findings, the therapeutic modalities tend to depend on the clinical symptoms, rather than the objective imaging findings.

MRI is a non-invasive and a very sensitive tool in detecting the early bony change such as bone marrow oedema, but it has some limitation in that it may have false positive or false negative results in the detection of the patella-femoral (PF) lesions. Bone scintigraphy is relatively sensitive because it reflects the early physiological changes of joints. But its image is planar that it cannot give enough information for the anatomic localization, and the image is overlapped.

To compensate for the defects of these imaging methods, bone single photon emission computed tomography (SPECT) has emerged as useful imaging tools in the diagnosis of OA.

Based upon the fact that subchondral bony changes precede joint space narrowing in OA, bone SPECT seems to be a very useful tool in early OA, reflecting the early bony changes.

The use of SPECT/CT offers the benefit of combined anatomical, mechanical (CT) and functional imaging (SPECT), which represents a relevant improvement in preoperative diagnosis and follow-up after procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient above 30 years old.
* Clinically diagnosed osteoarthritis before treatment.
* Patient with refractory active osteoarthritis (not responding to treatment).
* Ability to sleep in fixed position for about 25 minutes
* Ability to provide informed consent.

Exclusion Criteria:

* Patient with resolved osteoarthritis.
* patient with other disease in joints:

  * Avascular necrosis
  * Stress fracture
  * Neuropathic pain

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult patient above 30 years old.
  * Clinically diagnosed osteoarthritis before treatment.
  * Patient with refractory active osteoarthritis (not responding to treatment).
  * Ability to sleep in fixed position for about 25 minutes
  * Ability to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Detecting different pattern of osseous MDP uptake in patient with osteoarthritis in hip joints and/or knees in relation to clinical and simple radiographic findings. | Baseline
  Osteoarthritic patients will be examined with 99mTc-methylene diphosphonate (MDP) bone SPECT, the sites of uptake will be localized.
  Simple radiograph and physical examination will be assessed.The relationships between clinical findings, simple radiographic findings and the intensity of uptake in SPECT will be analyzed.